CLINICAL TRIAL: NCT04984187
Title: Effectiveness of High Intensity Laser Therapy Plus Therapeutic Interventions in Treatment of Girls Gymnasts With Non-specific Wrist Pain
Brief Title: Effect of High Intensity Laser Versus Plus Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hanaa 6
Record Dates: First submitted 2021-07-07; First posted 2021-07-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Effect of High Intensity Laser Plus Exercises on Wrist Pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser group (Other): High Intensity Laser Therapy only , this group will receive laser for 4 weeks three times /week
  Interventions: Device: high intensity laser only
- Exercise group (Other): Exercise , selected physiotherapy exercises will receive for 4 weeks ,3times/week
  Interventions: Other: exercise
- High intensity laser grouo (Experimental): High intensity laser plus exercise will receive the selected exercises and laser 4 weeks, 3 times/week
  Interventions: Other: high intensity laser plus exercise

INTERVENTIONS:
Other: high intensity laser plus exercise — high intensity laser plus exercise
  Arms: High intensity laser grouo
Device: high intensity laser only — high intensity laser only
  Arms: Laser group
Other: exercise — exercise only
  Other Names: exercise only
  Arms: Exercise group

SUMMARY:
High-intensity laser therapy (HILT) has been used more recently in the therapeutic protocols of musculoskeletal pain management. This study is conducted to find out the effect of high intensity laser therapy only versus high intensity laser pulse exercises on level of wrist pain, function and Joint position sense in girls Gymnasts

DETAILED DESCRIPTION:
Effect of high intensity laser plus exercises on wrist pain ..three groups of gymnastics girls suffer from non specific wrist is allocating ..the first group will receive exercises only , the second will receive laser only while the third will receive exercises plus laser

ELIGIBILITY:
Inclusion Criteria:

* All girls diagnosed with generalized chronic wrist pain and referred by orthopaedic physician.
* Their age between 10-16 years old
* They will be able to follow instructions.
* All are medically stable

Exclusion Criteria:

* • Bone fractures and tumors.

  * Cases after plastic surgery.
  * Hypertension (due to secondary vasoconstriction)
  * Diabetes mellitus
  * Pacemakers

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
PRWE | pre and post 4 weeks of intervention, decrease score indicate improvement
  The PRWE is a 15-item questionnaire that is used to rate wrist outcomes based on patient pain and function and is based on an 11-point (0-10) scale.

SECONDARY OUTCOMES:
JBS | pre and post 4 weeks of intervention, decrease score indicate improvement
  JPS assesses precision or accuracy in repositioning a joint at a predetermined target angle

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa Mohsen, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No